CLINICAL TRIAL: NCT03072485
Title: Phase 1 Study of the Effects of Combining Topical FDA-approved Drugs on Age-related Pathways on the Skin of Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Anne Chang (Other)
Responsible Party: Sponsor-Investigator, Anne Chang, Associate Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB-37203
Record Dates: First submitted 2017-02-27; First posted 2017-03-07 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Aging
Keywords: aging
MeSH Terms: interventions — Sirolimus; Metformin; Diclofenac

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sirolimus, metformin, diclofenac (Other): First five enrolled participants
  Interventions: Drug: Sirolimus; Drug: Metformin; Drug: Diclofenac
- Metformin, diclofenac (Other): Sixth to tenth enrolled participants
  Interventions: Drug: Metformin; Drug: Diclofenac

INTERVENTIONS:
Drug: Sirolimus — Topical sirolimus applied to the skin
  Arms: Sirolimus, metformin, diclofenac
Drug: Metformin — Topical metformin applied to the skin
Drug: Diclofenac — Topical diclofenac applied to the skin

SUMMARY:
This is a phase 1 study in healthy adult volunteers to examine the effects of 3 FDA approved medications on skin aging when applied in topical form. This is an open label, placebo controlled study.

DETAILED DESCRIPTION:
The primary endpoint of the study is the profile of differences in transcript levels of age-associated genes such as those in the lamin-A, insulin like growth factor (IGF) and NFKB pathways as well as noncoding RNAs in topical agent-exposed arm skin versus placebo exposed arm skin in healthy volunteers. The secondary endpoints include (1) differences in skin wrinkling using a 4 point Likert scale for wrinkle severity between placebo and topical agent exposed arm skin after 4 weeks of usage; (2) the type and severity of adverse events, both systemic and skin localized after exposure to both topical agent and placebo vehicle cream.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 55 years
2. Female
3. All 4 grandparents of European descent
4. Fitzpatrick Skin type 1-3 (fair skin type)
5. Presence of moderate to severe fine wrinkling on arm skin
6. Presence of moderate to severe dyspigmentation on arm skin
7. Normal or overweight body mass index

Exclusion Criteria:

1. History of laser treatment or chemical peels to to arm
2. History of topical anti-aging products (includes retinol, tretinoin, tazarotene, azelaic acid, hydroquinone) to skin within 6 weeks of starting study
3. History of surgical procedures to arm skin area including removal of benign or malignant skin cancers in the area of topical study agent application
4. Current skin conditions in the area of arms including seborrheic keratosis, rosacea, eczema that may obscure study assessment
5. History of abnormal scarring
6. Uncontrolled medical problems including concurrent infection or malignancy at time of enrollment
7. Unable to provide and sign written informed consent
8. Unable to comply with study-related procedures including keeping study diary, application of topical study agents, avoidance of direct sun exposure >5 minutes per day or ultraviolet tanning bed usage
9. Not willing to provide two small skin biopsies at end of study
10. Known allergy to sirolimus, diclofenac or metformin.
11. Known immunosuppression including organ transplant, HIV, autoimmune disease, and chronic leukemia or lymphoma
12. Fasting blood sugar above the upper limit of normal for Stanford laboratory
13. Diarrhea
14. Use of greater than one alcoholic beverage per day
15. Stress such as surgery or trauma within 2 weeks of enrollment
16. Liver disease such as hepatitis B or C
17. Planning to embark on dieting, caloric restriction or new exercise regimen during the study to lose weight.
18. Unable to refrain from using any topical agent on arms besides the study agents provided for duration of study.
19. Hematocrit, hemoglobin, platelets, white blood cell count, serum Na, K, Cr, aspartate aminotransferase (AST), alanine aminotransferase (ALT) greater or lesser than 1.5 times limits of normal.
20. History of heart failure, coronary artery disease, including angina, coronary artery bypass graft, pacemaker or stent placement
21. History of bleeding or ulcers of the gastrointestinal tract
22. History of diabetes mellitus
23. Current use of blood thinners (includes heparin, warfarin and aspirin)
24. Current use of strong cytochrome P 450 (CYP) 3A4 inhibitor and/or P-gp (examples include ketoconazole, voriconazole, itraconazole, erythromycin, clarithromycin) or strong inducers of CYP3A4 and/or P-gp (examples include rifampin or rifabutin)
25. Abnormal lipid panel as defined by upper limit of normal at Stanford laboratory

Min Age: 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-02-22 (Actual); Study Completion 2019-02-22 (Actual)

PRIMARY OUTCOMES:
Profile of gene transcript changes | 4 weeks
  Profile of gene transcript changes

SECONDARY OUTCOMES:
Wrinkle score | 4 weeks
  on Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Anne Chang, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Dermatology, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No